CLINICAL TRIAL: NCT05022524
Title: Exploring Novel Uses of Microbiota Therapy for Managing the Side Effects of Psychiatric Pharmaceutical Interventions: An N-of-1 Pilot and Feasibility Study
Brief Title: Exploring Novel Uses of Microbiota Therapy for Managing the Side Effects of Psychiatric Pharmaceutical Interventions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 119638
Record Dates: First submitted 2021-07-30; First posted 2021-08-26 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Depression, Anxiety
Keywords: Probiotics; Psychiatry; Weight
MeSH Terms: conditions — Depression; Anxiety Disorders; Body Weight | interventions — Acetates

STUDY DESIGN:
Intervention Model Description: N-of-1 type prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transition-Age Adults (Experimental): 16-25 year old patients on stable dose of antipsychotic medication for treatment of depression or anxiety.
  Interventions: Dietary Supplement: Acetate (Apple Cider Vinegar)

INTERVENTIONS:
Dietary Supplement: Acetate (Apple Cider Vinegar) — Consumer-grade apple cider vinegar (ACV) capsules will have extra enteric coating applied for delivery further into the GI tract.

SUMMARY:
To determine the feasibility of whether the addition of key prebiotics administered orally can mitigate some of the most problematic side-effects of the most common psychiatric medications - weight gain and metabolic abnormalities caused by some antidepressants, mood stabilizers and antipsychotics. In the initial part of the study, we aim to determine feasibility of the study and evaluate participant compliance.

Our clinical trial will encourage the growth of Akkermansia muciniphila (AM) through enteric-coated orally-administered acetate (apple cider vinegar powder in capsules) in 16-to-28 year-old patients who have already experienced weight gain while on stable doses of psychiatric medication, with the hypothesis that the addition of this prebiotic will result in alterations in gut microbiota and measurable weight loss, as well as improvement in metabolic measurements.

Primary Objective:

* To evaluate feasibility of using acetate in a large-scale clinical trial, including considerations for protocol, study agent, recruitment, retention, adverse events, budget, staff, facility, and patient experience
* To estimate effect size of change in AM relative abundance by measuring pre- and post-intervention levels for use in designing future large-scale clinical trials

Secondary Objectives:

* To determine whether acetate administered orally shows an observable effect on weight gain as a side effect from antidepressants, mood stabilizers, and/or antipsychotics in a sample of participants already on stable doses of at least one of these medications
* To determine changes in metabolic syndrome profile, as indicated by blood pressure and high-density lipoprotein.
* To conduct preliminary analyses on any possible changes in mood/anxiety symptoms pre- versus post-intervention
* To identify and define other potential confounders or effect modifiers of our primary and secondary objectives that should be considered in future study designs

ELIGIBILITY:
Inclusion Criteria:

For an eligible patient, all inclusion criteria must be answered "yes"

1. Signed informed consent obtained prior to any study-related activities
2. Patients of FEMAP who are between the ages of 16 and 28
3. Currently on a stable dose of an antidepressant, mood stabilizer, and/or antipsychotic drug AND have experienced what they deem to be problematic weight gain (approximately greater than 5% of initial body weight) that was temporally linked with initiating the drug, as confirmed by a psychiatrist
4. Have a body mass index of ≥ 21.7 kg/m2 (midpoint of normal BMI (18.5-24.9).

Exclusion Criteria:

1. Participants who are unable to follow multi-step instructions independently, as determined by the treating psychiatrist.
2. Participants who are pregnant or planning to get pregnant
3. Patients on medications that have weight loss as a potential side effect i.e. topiramate, metformin, psychostimulants.
4. Current active eating disorder i.e. bulimia nervosa, binge eating disorder, anorexia nervosa
5. Currently on a weight-loss diet plan i.e. ketogenic diet, detox diet
6. Currently using a medication for weight loss i.e. Contrave (bupropion / naltrexone), Saxenda (liraglutide)
7. Current use of dietary supplements for weight loss i.e. garcinia cambogia; or use within 4 weeks prior to study initiation
8. Bowel surgery
9. Crohn's disease or other bowel conditions
10. Blood/bleeding/liver/kidney disorders
11. Currently enrolled in other clinical trial which may affect their study outcome

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment success | 5 months
  Number of potential participants approached to number expressing interest, and number invited to number recruited (recruitment success)
Feasibility: Retention | 5 months
  Number recruited to number retained (attrition)
Feasibility: Adherence | 5 months
  Number adhering to intervention protocol quantified through number of capsules returned at end of trial
Feasibility: Adverse Events | 5 months
  A study-specific data form for collecting adverse events
Akkermansia Muciniphila abundance | 5 months
  Relative abundance (proportion) of AM in stool at inception compared to all other species identified, and change in relative abundance from pre- to post-intervention

SECONDARY OUTCOMES:
Body Weight | 5 months, recorded monthly
  Standard Medical-grade floor scale
Metabolic Indicator: Blood pressure | 5 months
  Blood pressure using medical-grade arm cuff (mm/Hg, Systolic and Diastolic)
Metabolic Indicator: High-Density Lipoproteins | 5 months
  HDL cholesterol assayed from antecubital blood draw, expressed in mg/dL
Mood: Depression | 5 months, captured monthly
  Quick Inventory of Depressive Symptomatology (QIDS-SR, Rush et al. 2003) - baseline scores to describe the sample, change from pre-post intervention to explore potential treatment effect
Mood: Anxiety | 5 months, captured monthly
  Overall Anxiety Severity and Impairment Scale (OASIS, Barlow et al. 2010) - baseline scores to describe the sample, change from pre-post intervention to explore potential treatment effect

CONTACTS AND LOCATIONS:
Locations (1):
- First Episode Mood and Anxiety Disorders Program (FEMAP), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers